CLINICAL TRIAL: NCT02777359
Title: Precutaneous High Risk Patent Foramen Ovale to Treat Migraine Headaches:A Prospective,Multicenter,Randomized,Controlled Trial
Brief Title: Precutaneous High Risk Patent Foramen Ovale to Treat Migraine Headaches
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other); Air Force Military Medical University, China (Other); Southwest Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2015-008
Record Dates: First submitted 2016-05-04; First posted 2016-05-19 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Patent Foramen Ovale
Keywords: patent foramen ovale; migraine; treatment
MeSH Terms: conditions — Foramen Ovale, Patent; Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- the closure group (Experimental): In the closure group, the transcatheter closure of PFO was performed using the made-in-China occluders approved by SFDA, in combination of clopidogrel(50mg/d, 3mon) and aspirin (0.1g/d, 6mon), i.e. oral administration of aspirin (0.1g/d) and clopidogrel (50mg/d) at 48h before the closure; the low molecular weight heparin (LMWH) was routinely given at 48h after the closure; and some pain-relief drugs could be temporarily administered in the patients with acute onset of migraine.
  Interventions: Procedure: the transcatheter closure of PFO
- the medication group (No Intervention): In the medication group, in combination of clopidogrel (50mg/d, 3mon) and aspirin (0.1g/d, 6mon), current medication resumed, including conventional prescription for migraine as β-receptor blockers, calcium-ion antagonists, antiepileptics, antidepressants and non-steroid anti-inflammatory drugs (NSAID).

INTERVENTIONS:
Procedure: the transcatheter closure of PFO — the transcatheter closure of PFO was performed using the made-in-China occluders approved by SFDA,clopidogrel(50mg/d, 3mon) , aspirin (0.1g/d, 6mon), i.e. oral administration of aspirin (0.1g/d) and clopidogrel (50mg/d) at 48h before the closure; the low molecular weight heparin (LMWH) was routinely given at 48h after the closure; and some pain-relief drugs could be temporarily administered in the patients with acute onset of migraine.
  Arms: the closure group

SUMMARY:
The foramen ovale, a kind of physiologic channel in the interatrial septum in the heart at embryonic stage, is closed normally at 5-7 months after birth. When it is not closed, it is referred to as the patent foramen ovale (PFO), which is found in approximately 1/4 of general population. It was shown in the studies in recent years that the risks of cryptogenic stroke, migraine, peripheral arterial embolism and decompression sickness in the patients with PFO were several times higher than those in healthy people. Therefore, PFO, previously considered a condition without the necessity of treatment, causes the attention of many experts and scholars around the world. Migraine with or without aura is defined as one of the most disabling chronic diseases, since according to WHO, the disability adjusted life year caused by migraine was second only to that by non-fatal stroke in 2005. In recent years, an increasing number of researches suggested that migraine is closely related to the right-to-left shunt (RLS) in the heart. And PFO is clinically considered as the most common cause of RLS.

The closure treatment for PFO-induced migraine has been gradually applied in several hospitals in China. The relationship of PFO with migraine, however, was not evaluated systematically based on specific standards, unfortunately leading to non-inclusion of many high-risk patients with PFO in the evaluation. The following aspects are to be fully recognized: the selecting and screening procedures for the high-risk population with PFO-induced migraine; the indications and standards of closure treatment for PFO in the patients with PFO-induced migraine; and the possibility that the made-in-China occluders substitute for those imported in the prevention from migraine. Furthermore, there is still a lack of prospective, multi-center, randomized and controlled studies in this subject, and standard or normal screening and treatment procedures have not yet been established in China. From this point, the investigators developed the Chinese people-specific procedures and standards of diagnosis of PFO-induced migraine in this study, based on current standards and methods of diagnosis, treatment and prevention of PFO-induced migraine in foreign countries. And the investigators prospectively adopted continuous inclusion of the high-risk patients with PFO-induced migraine, who were randomly divided into the closure treatment (transcatheter closure of PFO) group and the medication (drugs administered alone) group at the ratio of 1:1., in order to evaluate if the interventional treatment is better than the medication alone in these patients, to assess the efficacy and safety of the made-in-China occluders in the interventional treatment and prevention of PFO-induced migraine, and to identify the incidence of PFO in the patients with migraine in China and develop the Chinese people-specific screening protocols of PFO-induced migraine.

ELIGIBILITY:
Inclusion Criteria:

* migraine headaches with or without aura,migraine onset before age 50
* >3 migraine attacks or 5 migraine days per month
* failed ≥2 commonly accepted migraine medications:β-receptor blockers, calcium-ion antagonists, antidepressants and non-steroid anti-inflammatory drugs (NSAID).
* PFO documented by TTE or TEE
* PFO meet one of the following conditions:RLS in rest documented by cTTE or cTCD,combine with ASA,the primary patition mobility≥6.5mm,the diameter of PFO≥4mm, combine with Eustachian Valve or Chiari net.
* age 18-60
* else:independent in daily activities,to comply with complete follow-up experiment design

Exclusion Criteria:

* contraindication to antiplatelet or anticoagulant
* inferior vena cava or pelvic vein thrombogenesis leading to complete obstruction,systemic or local infection,septicemia,heart lumen thrombosis
* pregnancy
* combine with pulmonary hypertension or PFO made for a particular channel
* severe allergy to nickel

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
migraine days after randomization | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Yu Shun, PHD, Study Chair — First Affiliated Hospital of Xian JiaotongUniversity
Locations (1):
- First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Zhao E, Du Y, Xie H, Zhang Y. Modified Method of Contrast Transthoracic Echocardiography for the Diagnosis of Patent Foramen Ovale. Biomed Res Int. 2019 May 9;2019:9828539. doi: 10.1155/2019/9828539. eCollection 2019. PMID 31211145